CLINICAL TRIAL: NCT05667727
Title: The Effect of Adding Nebulized Epinephrine in Asthma Exacerbation Management in Pediatric Age Group Compared to Standard of Care: Superiority Trial
Brief Title: The Effect of Nebulized Epinephrine in Asthma Exacerbation in Pediatric Age Group With the Standard Treatment Compared to Standard Treatment Using Improvement PRAM Score as a Primary Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Adnan Juma Al Rawahi, Emergency Medicine Resident, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R2016
Record Dates: First submitted 2022-11-07; First posted 2022-12-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-04

CONDITIONS: Shortness of Breath; Asthma in Children; Epinephrine Causing Adverse Effects in Therapeutic Use; Salbutamol Adverse Reaction
MeSH Terms: conditions — Dyspnea | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: both groups will receive salbutamol and ipratropium as back to back nebulization for 3 times. Then the candidate will be randomized into experimental group (epinephrine nebulization) and the control group (salbutamol nebulization as 4th nebulization)
Who Masked: Participant, Care Provider, Investigator
Masking Description: the clinical pharmacist will label the medications according to coding system. 2 boxes will be available, one for weight less than 20kg and other box for patient weight more than or equal of 20 kg. Both boxes will contain both medications (epinephrine and salbutamol) in identical syringe with the same volume.
  The patient, physician and the nurse will be blinded to the 4th nebulization (experimental intervention)
  Once patient get enrolled in the study and received the standard of care (back to back nebulization), the nurse with take the experimental intervention according to the weight and the coding which been done the pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- epinephrine group (Experimental): this arm will include the participant who will receive back to back nebulization (standard of care) plus epinephrine nebulization.
  Interventions: Drug: nebulized epinephrine
- control group (Active Comparator): in this arm, participant will receive the standard of care treatment (salbutamol and ipratropium, back to back) plus salbutamol as 4th nebulization.
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: nebulized epinephrine — we are using 1:1000 epinephrine into nebulization form
  Arms: epinephrine group
Drug: Salbutamol — Patient will receive salbutamol as 4th nebulization.
  Other Names: The control
  Arms: control group

SUMMARY:
Our study aiming to look in improvement of Pediatric Respiratory Assessment Measure (PRAM) score as a primary outcome. The secondary outcomes involving the need for second step management, need for admission and possible side effects.

It's double blinded randomized control study comparing Nebulized Epinephrine with standard treatment (salbutamol + Ipratropium) versus the standard treatment only in pediatric patient.

A pilot study will be conducted before to detect the sample size required and data will be collected at deferent interval post treatment targeting intension to treat for analysis.

DETAILED DESCRIPTION:
Because there are no previous studies with the same methodology found, pilot study will be conducted to estimate the sample size.

Patients who are eligible to be enrolled in the study will be randomized into two group (after receiving the standard of care, 3 back to back nebulization (salbutamol and ipratropium bromide)) , the experimental group will be given epinephrine (1ml of 1:1000) as nebulization and the control group will receive salbutamol nebulization as 4th nebulization.

PRAM score with calculated before and at 60, 80, 100 min after the treatment.

ELIGIBILITY:
* Inclusion Criteria:

  * Pediatric age group 3 - 12 years
  * known to have asthma
  * Initial PRAM Score showed moderate to severe asthma exacerbation
* Exclusion Criteria:

  * History of lung or upper airway disease other than asthma:

    * bronchiolitis, anaphylaxis, pertussis, vocal cord dysfunction, foreign body aspiration, bronchopulmonary dysplasia, cystic fibrosis and lower airway mass effects
  * History of congenital heart disease or cardiac arrhythmia or heart failure.
  * Known hypertension
  * Impending respiratory failure (Decreasing mental status, Respiratory fatigue, Impending respiratory arrest, Hypoxemia (pO2 < 60 mmHg), pCO2 could be normal or high)
  * Allergy or hypersensitivity to epinephrine
  * Patient/Parents refusal to participate in the study

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
change in pediatric respiratory assessment measure (PRAM) score | at (60) mints
  treating physician will calculate the PRAM score before and immediately after the intervention by 20 mins, if there is no change in PRAM score or the case worsen, candidate will receive further treatment, but if he/she improved, will be assessed in the second interval.
change in pediatric respiratory assessment measure (PRAM) score | at (80) mints
  immediately after the intervention by 40 mins, candidate will be assessed, calculating the PRAM score again, and decide he/she will need further treatment or to continue observation.
change in pediatric respiratory assessment measure (PRAM) score | at (100) mints
  immediately after the intervention by 90 mins, candidate will be assessed again, calculating the PRAM score and decide about if he will need further treatment or no.
  Total observation will be almost 2 hours in order to look for other outcome as well.

SECONDARY OUTCOMES:
Emergency Department (ED) length of stay | from the randomization up to 4 hours
  "during the assessment", after the exposure
  This outcome will be decided upon each reassessment intervals, at any time during assessment if there is no change in PRAM score or worsening patient will receive further treatment as decided before and his enrollment in the study will be ended here.
The rate for admission | from the randomization up to 4 hours
  "during the assessment"
  this will be determined at the disposal plan for each candidate from the emergency department, either admission or discharge home.
rate of any side effect of nebulized epinephrine | from the randomization up to 4 hours
  "during the assessment"
  Each candidate will be assessed throughout the enrolment in the study, starting from the administration of the medication till 2 hours post exposure.
The need for respiratory support (O2, Non-invasive ventilation, intubation) | from the randomization to the disposal time
  "during assessment"
The rate of revisit to Emergency Department within 72 hours of the index visit | Till 72 hours post discharge
  "after discharge"

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hospital, Muscat, Oman